CLINICAL TRIAL: NCT03857659
Title: Serial Third Trimester Abdominal Circumference and Amniotic Fluid Measurements Versus Routine Care: A Randomized Controlled Trial (STAR Trial)
Brief Title: Serial Third Trimester Abdominal Circumference and Amniotic Fluid Measurements Versus Routine Care
Acronym: STAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID related termination
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-18-1074
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Fetal Growth Abnormality; Amniotic Fluid; Disorder
Keywords: Pregnancy; Ultrasound; neonatal morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Point of care ultrasound (POC-US) (Experimental): Point of care ultrasound (POC-US) to measure abdominal circumference and amniotic fluid every 4 weeks from 28-36 weeks
  Interventions: Diagnostic Test: Point-of-care ultrasound (POC-US); Diagnostic Test: Formal ultrasound
- Routine antenatal care (Active Comparator): Routine care with fundal height measurement at each antenatal appointment every 2 weeks from 28-36 weeks. As well as clinically indicated obstetric ultrasound by a Registered Diagnostic Medical Sonographer (RDMS)
  Interventions: Diagnostic Test: Routine antenatal care; Diagnostic Test: Formal ultrasound

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound (POC-US) — POC-US evaluation will be conducted using the portable ultrasound machine, which is capable of straight-line measurements for assessment of the amniotic fluid, as well as ellipse measurements for determination of abdominal circumference. POC-US evaluation will be conducted every 4 weeks from 28-36 weeks.
  Arms: Point of care ultrasound (POC-US)
Diagnostic Test: Routine antenatal care — Routine care with fundal height measurement at each antenatal appointment every 2 weeks from 28-36 weeks. As well as clinically indicated obstetric ultrasound by a Registered Diagnostic Medical Sonographer (RDMS)
  Arms: Routine antenatal care
Diagnostic Test: Formal ultrasound — Formal growth ultrasound performed between 36-38.6 weeks by RDMS.

SUMMARY:
The purpose of this study us to compare the rate of prenatal identification of abnormal fetal growth or amniotic fluid between clinical evaluation of uterine size by symphysis fundal height (SFH) measurements versus point-of-care ultrasound (POC-US) evaluation of abdominal circumference (AC) and maximum vertical pocket (MVP).

ELIGIBILITY:
Inclusion Criteria:

* Maternal age of 18 at the time of consent
* Singleton gestation
* Ultrasound examination that confirms or revises the estimated date of delivery (EDD) before 22 0/7 weeks of gestational age
* Gestational age ≥ 24 weeks gestation

Exclusion Criteria:

* Abnormal aneuploidy screening (1st trimester screening, 2nd trimester screening, integrated screening, NIPT)
* Fetal chromosomal or genetic abnormalities
* Fetal malformations or soft markers identified on fetal anatomy survey
* Current pregnancy is a result of in vitro fertilization
* Documented uterine bleeding after 24 weeks gestation. Unobserved self-reported bleeding with confirmed intact pregnancy on ultrasound after the bleeding episode is not an exclusion criterion.
* Uterine/placental abnormalities including uterine malformations (i.e bicornuate uterus, didelphus uterus), abnormal placentation (placenta previa, accrete, percreta), uterine fibroids.
* Cerclage in the current pregnancy
* History of intrauterine fetal demise
* Fetal isoimmunization or alloimmunization
* History of medical complications such as:

  * Cancer (including melanoma but excluding other skin cancers)
  * Endocrine disease including thyroid disease (recently diagnosed or whose medication dose is not stable), adrenal disease, diabetes mellitus (pregestational and gestational).
  * Renal disease with altered renal function (creatinine > 0.9 or proteinuria)
  * Epilepsy or other seizure disorder
  * Any collagen disease (lupus erythematosus, scleroderma, etc.)
  * Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes)
  * Hematological disorder including alloimmune and isoimmune thrombocytopenia but excluding mild iron deficiency anemia (Hb > 9 gm/dl). Patients with sickle cell disease are excluded.
  * Chronic pulmonary disease including asthma requiring regular use of medication and active tuberculosis (TB). An asthma inhaler used on an as needed basis (PRN) for a cold or an asthma attack is not considered regular use.
  * Heart disease except mitral value prolapse not requiring medication
  * Cardiovascular disorders: chronic hypertension
  * Liver disorders accounting for cholestasis
  * Infectious diseases: HIV, Cytomegalovirus (CMV), toxoplasmosis, parvovirus B19

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 36 weeks GA
  Abnormal fetal growth or amniotic fluid as assessed by clinical evaluation of uterine size by SFH versus POC-US evaluation.
Number of participants with abnormal fetal growth or amniotic fluid | From 36 weeks Gestational age (GA) to 38.6 weeks GA
  Abnormal fetal growth or amniotic fluid as assessed by formal ultrasound by RDMS

SECONDARY OUTCOMES:
Sensitivity of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
Sensitivity of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
Specificity of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
Specificity of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
Positive predictive value of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
Positive predictive value of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
Negative predictive value of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
Negative predictive value of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
False positive rate of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
False positive rate of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
False negative rate of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
False negative rate of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
Positive likelihood ratio of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
Positive likelihood ratio of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
Negative likelihood ratio of diagnostic methods for identification of abnormal fetal growth or amniotic fluid | From 28 weeks Gestational age (GA) to 38.6 weeks GA
  Test performance characteristics of SFH measurements and POC US for identification of abnormal fetal growth or amniotic fluid using formal USE as the diagnostic standard.
Negative likelihood ratio of diagnostic methods for identification of birthweight < 10th percentile or > 90th percentile | From 28 weeks Gestational age (GA) to time of delivery
  Test performance characteristics of SFH measurements and POC US for identification of birthweight < 10th percentile or > 90th percentile using the neonates' gestational age at delivery as the standard
Number of referrals for formal USE. | From 28 weeks Gestational age (GA) to 36 weeks GA
Number of participants with composite neonatal morbidity | at delivery
  Composite neonatal morbidity is defined as any of the following:
  * 1) Apgar score < 3 at 5 min, 2) birth trauma, 3) hypotension requiring vasopressor support, 4) hypoxic-ischemic encephalopathy, 5) infection, 6) intracranial or subgaleal hemorrhage, 7) meconium aspiration syndrome, 8) perinatal death, 9) respiratory support, or 10) seizure.
    4. The rate of composite neonatal morbidity, including any of the following:
  * 1) Apgar score < 3 at 5 min, 2) birth trauma, 3) hypotension requiring vasopressor support, 4) hypoxic-ischemic encephalopathy, 5) infection, 6) intracranial or subgaleal hemorrhage, 7) meconium aspiration syndrome, 8) perinatal death, 9) respiratory support, or 10) seizure.
Number of participants with composite maternal morbidity | labor until delivery (total time is about 1-48 hrs)
  Composite maternal morbidity is defined as any of the following:
  o 1) chorioamnionitis, 2) cesarean delivery in labor, 3) wound infection, 4) transfusion, 5) deep venous thrombus or pulmonary embolism, 6) admission to intensive care unit, 7) postpartum hemorrhage, or 8) death
Total costs of care from the health system perspective | from time of randomization until discharge (total time is about 15 weeks)
  6. The total costs of care from the health system perspective during the study period (from the date of enrollment through the mothers' post-delivery discharge and the infants' post-birth discharge). The hospital costs (for ER visits, admissions, delivery, and neonatal care) will be obtained from the Memorial Hermann Hospital cost-accounting system. The costs of physician services received during the study period by the mothers and the newborns will be estimated using relative value units (RVUs) based on claims data. The intervention arm will be augmented by the cost of the POC-US examinations. The POC-US costs will include the costs of the POC provider time (estimated based on limited time-motion studies, salary, and fringe data) and the depreciation costs of the portable ultrasound equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bicocca, MD, Principal Investigator — University of Texas Health Science Center of Houston
Locations (1):
- University of Texas Health Science Center of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No